CLINICAL TRIAL: NCT06940310
Title: Effects of Different Methods of Prescription and Monitoring of Resistance Training Intensity on Muscle Strength, Body Composition, and Psychological Well-being in Survivors of Breast Cancer
Brief Title: Different Resistance Training Intensity Prescription and Monitoring Methodologies: Effects on Strength, Body Composition, and Well-being in Survivors of Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Patronato Municipal de Deportes de Almería, Spain (Unknown)
Responsible Party: Principal Investigator, Alberto Soriano-Maldonado, PhD, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EFICAN/04/2025
Record Dates: First submitted 2025-03-28; First posted 2025-04-23 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: resistance training; muscular strength; health-related quality of life; exercise intensity; breast malignancy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Daily load-velocity-based training intensity adjustment (Experimental): At the beginning of the training session, the one-repetition maximum (1RM) will be estimated based on the individual's load-velocity relationship, using the general velocity associated with the 1RM for the exercises included in the session. Additionally, during the training sessions, intensity will be monitored, and load will be adjusted in real time by movement velocity.
  Interventions: Behavioral: Daily load-velocity-based training intensity adjustment.
- Training intensity prescription based on an initial 1RM estimation using load-velocity relationship. (Experimental): In the first training session, the one-repetition maximum (1RM) will be estimated based on the individual's load-velocity relationship, using the general velocity associated with the 1RM for the exercises included in the session. This 1RM will be used to prescribe exercise intensity throughout the intervention.
  Interventions: Behavioral: Training intensity prescription based on an initial 1RM estimation using load-velocity relationship
- Traditional training with intensity prescription based on 1RM testing. (Experimental): The traditional training group will follow a training program using the traditionally employed methodology for assessing and prescribing training intensity in breast cancer survivors. This methodology is based on an initial 1RM estimation conducted through a 1RM test, which will be used to prescribe the training load throughout the intervention.
  Interventions: Behavioral: Traditional training with intensity prescription based on 1RM testing.

INTERVENTIONS:
Behavioral: Daily load-velocity-based training intensity adjustment. — At the beginning of the training session, the one-repetition maximum (1RM) will be estimated based on the individual's load-velocity relationship, using the general velocity associated with the 1RM for the exercises included in the session. Additionally, during the training sessions, intensity will be monitored, and load will be adjusted in real time by movement velocity.
  Arms: Daily load-velocity-based training intensity adjustment
Behavioral: Training intensity prescription based on an initial 1RM estimation using load-velocity relationship — In the first training session, the one-repetition maximum (1RM) will be estimated based on the individual's load-velocity relationship, using the general velocity associated with the 1RM for the exercises included in the session. This 1RM will be used to prescribe exercise intensity throughout the intervention.
  Arms: Training intensity prescription based on an initial 1RM estimation using load-velocity relationship.
Behavioral: Traditional training with intensity prescription based on 1RM testing. — The traditional training group will follow a training program using the traditionally employed methodology for assessing and prescribing training intensity in breast cancer survivors. This methodology is based on an initial 1RM estimation conducted through a 1RM test, which will be used to prescribe the training load throughout the intervention.
  Arms: Traditional training with intensity prescription based on 1RM testing.

SUMMARY:
The goal of this clinical trial is to compare the effects of three different methods of prescribing and monitoring resistance training intensity on muscle strength, body composition, quality of life, fatigue, anxiety, and depression in breast cancer survivors.

DETAILED DESCRIPTION:
Breast cancer survival rates have significantly increased in recent years, highlighting the importance of effective interventions to address the long-term consequences of cancer and its treatments. Breast cancer survivors often experience muscle weakness, changes in body composition, fatigue, and psychological distress, which can negatively impact their quality of life. Resistance training has been widely recognized as a safe and effective strategy to counteract these effects, improving muscle strength, body composition, and psychological well-being.

Despite its benefits, the optimal method for prescribing and monitoring resistance training intensity in breast cancer survivors remains unclear. Traditional methods based on one-repetition maximum (1RM) testing may not fully account for individual variations in fatigue and performance. Alternative approaches, such as load-velocity relationships, allow for more precise and real-time adjustments to training intensity, potentially optimizing outcomes.

This randomized controlled trial aims to compare the effects of three different methods of resistance training intensity prescription and monitoring on muscle strength, body composition, quality of life, fatigue, anxiety, and depression in breast cancer survivors. The findings will contribute to developing evidence-based exercise guidelines, enhancing rehabilitation strategies and overall well-being in this population.

ELIGIBILITY:
Inclusion Criteria:

* To be >18 years old.
* To have a breast cancer diagnosis.
* To have finished chemotherapy, radiotherapy and/or surgery up to 10 years prior to the beginning of the study.

Exclusion Criteria:

* To present metastatic breast cancer.
* To have a planned surgery for breast reconstruction within three months after the start of the study.
* To present any absolute contraindication for exercising.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Muscular strength | Change from baseline to week 8
  The main variable of the present study will be muscle strength, assessed by determining peak isometric strength in the bench press and squat exercises using force platforms.

SECONDARY OUTCOMES:
Handgrip strength | Change from baseline to week 8
  Handgrip strength will be determined using a digital dynamometer (Model T.K.K.540; Takei Scientific Instruments Co, Ltd).
Muscle function (5STS) | Change from baseline to week 8
  Muscle function will be assessed using the 30-second sit-to-stand test. Additionally, the five-repetition sit-to-stand (5STS) test will be performed on force platforms, and the peak force of all repetitions will be recorded.
Height (scale) | Baseline
  Height will be determined using a scale (cm)
Body weight (InBody 770) | Change from baseline to week 8
  Body wieght (kg) will be determined using bioelectrical impedance analysis (InBody 770; InBody Co Ltd, Seoul, Korea).
Total fat mass (InBody 770) | Change from baseline to week 8
  Total fat mass (kg) will be determined using bioelectrical impedance analysis (InBody 770; InBody Co Ltd, Seoul, Korea).
Fat percentage (InBody 770) | Change from baseline to week 8
  body fat percentage (%) will be determined using bioelectrical impedance analysis (InBody 770; InBody Co Ltd, Seoul, Korea).
Fat-free mass (InBody) | Change from baseline to week 8
  Fat-free mass (kg) will be determined using bioelectrical impedance analysis (InBody 770; InBody Co Ltd, Seoul, Korea).
Visceral fat mass level (InBody) | Change from baseline to week 8
  Visceral fat mass level (U) will be determined using bioelectrical impedance analysis (InBody 770; InBody Co Ltd, Seoul, Korea).
Health-related quality of life (FACT-B) | Change from baseline to week 8
  Quality of life will be assessed using the Functional Assessment of Cancer Therapy-Breast (FACT-B) questionnaire. The global score ranges from 0 to 148 where higher scores indicate better quality of life.
Cancer-related fatigue (FACIT-F) | Change from baseline to week 8
  Fatigue will be assessed using the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) questionnaire. The score ranges from 0 to 52, where higher scores indicate lower levels of fatigue.
Anxiety and depression (HADS) | Change from baseline to week 8
  Anxiety and depression will be determined using the Hospital Anxiety and Depression Scale (HADS). Scores range from 0 to 21 for both HADS-A (Anxiety) and HADS-D (Depression) subscales, where higher scores indicate more severe symptoms of anxiety or depression.
Patient global impression of change | Week 8
  Patient global impression of change after the intervention will be evaluated at the end of the trial using a single Likert-type question.

OTHER OUTCOMES:
Rate of perceived exertion (RPE) | Through intervention completion, during 8 weeks. From day 1 to day 24.
  The rate of perceived exertion during the whole training session will be assessed at the end of each of the 24 intervention session using the modified Borg Scale (0-10) where higher scores mean higher perceived exertion.
Mood (Feeling Scale) | Through intervention completion, during 8 weeks. From day 1 to day 24.
  The mood perceived by the participants at the end of the session will be measured at the end of each of the 24 intervention session using the Feeling Scale. The scale ranges from -5 to 5, where higher scores indicate positive affect toward physical activity.
Perceived fatigue (VAS-F) | Through intervention completion, during 8 weeks. From day 1 to day 24.
  The fatigue perceived by the participants at the end of the session will be assessed at the end of each of the 24 intervention session using a visual analog scale for fatigue (VAS-F). The scale ranges from 0 to 10, where higher scores indicate greater fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Soriano-Maldonado, Principal Investigator — Universidad de Almeria
Locations (1):
- University of Almeria, Almería, Almeria, Spain

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data will be shared once the study is finalized and the main results are published. IPD can be obtained by contacting the responsible party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: One year (12 months) after study completion and once the results have been published.
Access Criteria: The PI must be contacted and a consensus must be reached on potential co-authorship.